CLINICAL TRIAL: NCT00106496
Title: A Multi-Center Study to Assess the Impact of Topical Corticosteroids on the Safety and Efficacy of Protopic Ointment in the Short-Term Treatment of Atopic Dermatitis and to Assess Protopic in the Long-term Management of Atopic Dermatitis
Brief Title: A Multi-Center Study of Short and Long-term Use of Protopic Ointment in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-04-002
Record Dates: First submitted 2005-03-25; First posted 2005-03-28 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Dermatitis, Atopic
Keywords: Treatment Effectiveness; Treatment Efficacy; Immunomodulator, Topical; Tacrolimus, Topical; Dermatitis, Atopic; Eczema, Atopic; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1A (Experimental)
  Interventions: Drug: Protopic
- 1B (Active Comparator)
  Interventions: Drug: Corticosteroid
- 2 (Experimental): Open label
  Interventions: Drug: Protopic
- 3A (Experimental)
  Interventions: Drug: Protopic
- 3B (Placebo Comparator)
  Interventions: Drug: placebo
- 4 (Experimental): Open label
  Interventions: Drug: Protopic

INTERVENTIONS:
Drug: Protopic — topical
  Other Names: tacrolimus ointment; FK506 ointment
  Arms: 1A; 2; 3A; 4
Drug: Corticosteroid — topical
  Arms: 1B
Drug: placebo — topical
  Arms: 3B

SUMMARY:
The purpose of the study is to determine the impact of topical corticosteroids on the safety and effectiveness of Protopic Ointment in the short-term treatment of moderate to severe Atopic Dermatitis and to compare the safety and effectiveness of Protopic Ointment to placebo in the long-term management of Atopic Dermatitis

DETAILED DESCRIPTION:
Study includes an interim short-term, open label period. Patients could also receive a second course of open label treatment dependent on disease exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have Atopic Dermatitis
* Patient must be at least 2 years of age

Exclusion Criteria:

* Patient is pregnant or breast feeding an infant

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2004-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
percentage of patients reporting cutaneous adverse events during the first 2 weeks of treatment | 2 weeks

SECONDARY OUTCOMES:
Percentage of patients reporting cutaneous adverse events overall | Day 4 through end of study

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (22):
- United States (22):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Irvine, California
  - Investigational Site, Loma Linda, California
  - Investigational Site, San Diego, California
  - New Haven, Connecticut
  - Miami, Florida
  - Investigational Site, Atlanta, Georgia
  - Investigational Site, Chicago, Illinois
  - Chicago, Illinois
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Investigational Site, Ann Arbor, Michigan
  - Investigational Site, Detroit, Michigan
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Lebanon, New Hampshire
  - Investigational Site, New York, New York
  - Investigational Site, Winston-Salem, North Carolina
  - Investigational Site, Cincinnati, Ohio
  - Investigational Site, Portland, Oregon
  - Investigational Site, Philadelphia, Pennsylvania
  - Investigational Site, Nashville, Tennessee
  - Investigational Site, Dallas, Texas

REFERENCES:
- [Background] Breneman D, Fleischer AB Jr, Abramovits W, Zeichner J, Gold MH, Kirsner RS, Shull TF, Crowe AW, Jaracz E, Hanifin JM; Tacrolimus Ointment Study Group. Intermittent therapy for flare prevention and long-term disease control in stabilized atopic dermatitis: a randomized comparison of 3-times-weekly applications of tacrolimus ointment versus vehicle. J Am Acad Dermatol. 2008 Jun;58(6):990-9. doi: 10.1016/j.jaad.2008.02.008. Epub 2008 Mar 21. PMID 18359127
- [Background] Paller AS, Eichenfield LF, Kirsner RS, Shull T, Jaracz E, Simpson EL; US Tacrolimus Ointment Study Group. Three times weekly tacrolimus ointment reduces relapse in stabilized atopic dermatitis: a new paradigm for use. Pediatrics. 2008 Dec;122(6):e1210-8. doi: 10.1542/peds.2008-1343. Epub 2008 Nov 17. PMID 19015204